CLINICAL TRIAL: NCT03844360
Title: Dose Individualization of Antineoplastic Drugs and Anti-Infective Drug in Children With Hematoplastic Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wei Zhao (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Antineoplastic Drugs001
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2019-04

CONDITIONS: Hematological Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Bortezomib; eltrombopag; Imatinib Mesylate; Dasatinib; pegaspargase; Anti-Infective Agents; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Antineoplastic Drugs and Anti-infective Drugs (Experimental): Bortezomib;eltrombopag;imatinib;dasatinib, pegaspargase and anti-infective drugs administered at standard dose for children with hematological neoplasms.
  Interventions: Drug: Bortezomib; Drug: Eltrombopag; Drug: Imatinib; Drug: dasatinib; Drug: Pegaspargase; Drug: Anti-Infective Drugs; Drug: PEGylated Recombinant Human Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Bortezomib — bortezomib was administered follow the doctor's advice.
  Other Names: Velcade
Drug: Eltrombopag — eltrombopag was administered follow the doctor's advice.
  Other Names: promacta
Drug: Imatinib — imatinib was administered follow the doctor's advice.
  Other Names: Gleevec
Drug: dasatinib — dasatinib was administered follow the doctor's advice.
  Other Names: sprycel
Drug: Pegaspargase — pegaspargase was administered follow the doctor's advice.
  Other Names: Oncaspar
Drug: Anti-Infective Drugs — anti-infective drugs was administered follow the doctor's advice.
Drug: PEGylated Recombinant Human Granulocyte Colony-Stimulating Factor — pegaspargase was administered follow the doctor's advice.
  Other Names: PEG-rhG-CSF

SUMMARY:
The investigators' purpose was to assess the feasibility of dosage individualization of the commonly used antineoplastic drugs and anti-infective drugs in children with hematoplastic disease.

DETAILED DESCRIPTION:
The investigators' purpose was to assess the feasibility of dosage individualization of the commonly used antineoplastic drugs and anti-infective drugs based on the opportunistic sampling strategy in children with confirmed or suspected hematological neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with hematological neoplasms
* Antineoplastic drugs or anti-infective drugs used as part of regular treatment

Exclusion Criteria:

* expected survival time less than the treatment cycle;
* patients with other factors that researcher considers unsuitable for inclusion.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change of plasma concentration of bortezomib | at(0-0.5)h,(0.5-3)h,(24-48)h,(48-72)h hours after administration
  To detect the plasma concentrations of bortezomib after administration
change of plasma concentration of eltrombopag | at (0.5-3)h,(3-6)h,(10-14)h,(20-24)h hours after oral administration
  To detect the plasma concentrations of eltrombopag after administration
change of plasma concentration of imatinib | at (0.5-2)h,(2-4)h,(10-14)h,(20-24)h hours after oral administration
  To detect the plasma concentrations of imatinib after administration
change of plasma concentration of dasatinib | at(0-0.5)h,(0.5-3)h,(10-14)h,(20-24)h hours after oral administration
  To detect the plasma concentrations of dasatinib after administration
change of plasma concentration of pegaspargase | at Day-1,Day(0-1),Day(3-5),Day(8-10),Day(13-14) after administration
  To detect the plasma concentrations of pegaspargase after administration
plasma concentration of anti-infective drug | through study completion, an average of 14 days
  To detect the plasma concentrations of anti-infective drug after administration

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (2):
- China (2):
  - Department of Pediatrics, the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - State Key Laboratory of Experimental Haematology, Department of Paediatric Haematology, Institute of Haematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tanjin, Tianjin Municipality

REFERENCES:
- [Derived] Zhang W, Chang LX, Zhao BB, Zheng Y, Shan DD, Tang BH, Yang F, Zhou Y, Hao GX, Zhang YH, van den Anker J, Zhu XF, Zhang L, Zhao W. Efficacy, Safety, and Population Pharmacokinetics of Eltrombopag in Children with Different Severities of Aplastic Anemia. J Clin Pharmacol. 2024 Aug;64(8):932-943. doi: 10.1002/jcph.2430. Epub 2024 Mar 18. PMID 38497347
- [Derived] Yang F, Zhang L, Zhao BB, Zhang JL, Liu XT, Li X, Tang BH, Zhou Y, Yang XM, van den Anker J, Zhu XF, Zhao W. Population Pharmacokinetics and Safety of Dasatinib in Chinese Children with Core-Binding Factor Acute Myeloid Leukemia. Clin Pharmacokinet. 2022 Jan;61(1):71-81. doi: 10.1007/s40262-021-01054-6. Epub 2021 Jul 9. PMID 34240339